CLINICAL TRIAL: NCT00851357
Title: The Efficacy of Telephone Counseling and the Centralized Distribution of Nicotine Replacement Therapy Through a Smoking Cessation Quitline
Brief Title: Telephone Counseling and the Distribution of Nicotine Patches to Smokers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: California Department of Health Services (Other)
Responsible Party: Principal Investigator, Shu-Hong Zhu, Professor, University of California, San Diego
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CDPH 05-45834
Record Dates: First submitted 2009-02-24; First posted 2009-02-25 (Estimated); Results first posted 2020-02-10 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Smoking Cessation
Keywords: Nicotine Replacement Therapy; Nicotine Patch; Smoking cessation; Telephone; Tobacco cessation; Counseling; Nicotine; Self-Help; Smoking abstinence; Tobacco Use Disorder
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Cessation; Tobacco Use Disorder | interventions — Tobacco Use Cessation Devices; Nicotine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Active patches and telephone counseling (Experimental): Proactive Telephone Counseling and 8-weeks of nicotine patches
  Interventions: Drug: Nicotine Patch; Behavioral: Telephone Counseling
- Placebo patches and telephone counseling (Placebo Comparator): Proactive Telephone Counseling and 8-weeks of placebo patches
  Interventions: Behavioral: Telephone Counseling; Drug: Placebo
- Telephone counseling (Active Comparator): Proactive Telephone Counseling
  Interventions: Behavioral: Telephone Counseling
- Active patches and materials (Active Comparator): 8-weeks of nicotine patches and materials
  Interventions: Drug: Nicotine Patch; Other: Self-Help Materials
- Placebo patches and materials (Active Comparator): 8-weeks placebo patches and materials
  Interventions: Drug: Placebo; Other: Self-Help Materials
- Materials (Active Comparator): Self-help materials
  Interventions: Other: Self-Help Materials

INTERVENTIONS:
Drug: Nicotine Patch — Subjects are randomized into 1 of 3 conditions: active, placebo or usual care. Usual care subjects are not mailed patches; however, we facilitate their use by providing a certificate that can be used by the State Medicaid program and some insurance companies to obtain free patches. For those mailed patches directly, we will mail 8 weeks of patches. Dosage depends on the number of cigarettes per day (cpd). Light smokers (6-10 cpd) will receive 6 weeks of 14 mg and 2 weeks of 7 mg patches. Heavy smokers (11+ cpd) will receive 4 weeks of 21 mg, 2 weeks of 14 mg and 2 weeks of 7 mg patches. Placebo patches will have no nicotine, but will be packaged to mimic the active patches.
  Other Names: Habitrol
  Arms: Active patches and materials; Active patches and telephone counseling
Behavioral: Telephone Counseling — Subjects call the Helpline and are screened for services. Eligible clients who give consent will be randomly assigned to a group.
  Subjects will be randomized into one of 2 behavioral conditions: telephone counseling or self-help materials. Telephone counseling includes a comprehensive pre-quit session (to include motivation, planning, and setting of a quit date and discussion of nicotine patch use) plus up to 5 proactive follow-up calls. Telephone counseling has several distinguishing features, namely proactive follow up counseling calls, a manualized protocol, and relapse-sensitive scheduling.
  Arms: Active patches and telephone counseling; Placebo patches and telephone counseling; Telephone counseling
Drug: Placebo — Placebo nicotine patch
  Other Names: Non-nicotine patch
  Arms: Placebo patches and materials; Placebo patches and telephone counseling
Other: Self-Help Materials — Subjects call the Helpline and are screened for services. Eligible clients who give consent will be randomly assigned to a group.
  Subjects will be randomized into one of 2 behavioral conditions: telephone counseling or self-help materials. Reading materials and written consent will be mailed to all study subjects the next business day.
  Arms: Active patches and materials; Materials; Placebo patches and materials

SUMMARY:
The primary purpose of this study is to determine the effects of distributing free nicotine replacement therapy (NRT) to tobacco quitline callers directly. Specifically, this study aims to:

1. Test if sending active nicotine patches directly will lead to a higher quit rate, compared to a condition where the quitline assists the smokers to obtain patches by other means (e.g. via their health plans).
2. Test if sending placebo patches directly will also lead to a higher quit rate.
3. Test if quitline counseling increases the quit rate when the smokers already receive the nicotine patches.

DETAILED DESCRIPTION:
Studies have shown that statewide tobacco quitlines can dramatically increase call volume by offering direct mailings of free nicotine replacement therapy (NRT) products. Sending free NRT such as patches to quitline callers, however, often requires a large budget because quitlines have a large number of smokers calling for help each year. A strong rationale is needed for state funding agencies to pay for the patches, which are generally considered the responsibility of health plans. This study will contrast the condition of sending nicotine patches directly from the quitline with a condition where the quitline assists smokers to obtain patches by other means, primarily through their health plans. The study aims to demonstrate that sending patches immediately after smokers call the quitline has a motivational effect that will lead to a higher quit rate than if smokers have to obtain the patches themselves, even if they are able to obtain them for free. To tease apart how much of the effect of sending patches directly from the quitline is due to the active ingredient in the patches and how much is due to motivational effects, this study adds a placebo condition. We hypothesize that the active patches condition will outperform the placebo condition, and the sending of placebo patches will outperform the condition in which the smokers obtain the nicotine patches themselves. We also hypothesize that counseling has its own effect on quitting above and beyond that of the nicotine patches. This study will supply data that can be used to decide what role nicotine replacement therapy should play in publicly funded tobacco cessation programs. Results will also add to the theoretical understanding of behavior change from which new, effective interventions can spring.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 years old
* Daily smoker
* >=6 cigarettes per day
* Ready to quit within one month
* First time quitline caller
* Valid phone number
* Valid address (no P.O. boxes)
* California resident
* Agree to participate in study and evaluation
* English or Spanish speaking

Exclusion Criteria:

* Uses other form of tobacco
* Use of Zyban or Chantix
* One of the following conditions: Severe allergy to adhesive tape, Arrhythmia, Angina, Heart attack within last year, Stroke within last year, Uncontrolled high blood pressure, Insulin-dependent diabetes, Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4200 (Actual)
Dates: Start 2009-02; Primary Completion 2010-10 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Hong Zhu, Ph.D., Principal Investigator — University of California, San Diego
Locations (1):
- University of Californian, San Diego: California Smokers' Helpline, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual Care: Subjects are not mailed nicotine patches; however, we facilitate their use by providing a certificate that can be used by the State Medicaid program and some insurance companies to obtain free patches.
- Patch (Placebo): Subjects are mailed patches directly, we will mail 8 weeks of patches. Dosage depends on the number of cigarettes per day (cpd). Light smokers (6-10 cpd) will receive 6 weeks of 14 mg and 2 weeks of 7 mg patches. Heavy smokers (11+ cpd) will receive 4 weeks of 21 mg, 2 weeks of 14 mg and 2 weeks of 7 mg patches. Placebo patches will have no nicotine, but will be packaged to mimic the active patches.
- Patch (Real): Subjects are mailed patches directly, we will mail 8 weeks of patches. Dosage depends on the number of cigarettes per day (cpd). Light smokers (6-10 cpd) will receive 6 weeks of 14 mg and 2 weeks of 7 mg patches. Heavy smokers (11+ cpd) will receive 4 weeks of 21 mg, 2 weeks of 14 mg and 2 weeks of 7 mg patches.
Period: Overall Study
Arm/Group | Usual Care | Patch (Placebo) | Patch (Real)
Started | 1200 | 1201 | 1799
Completed | 1200 | 1201 | 1799
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Patch (Placebo) | Patch (Real) | Total
Number analyzed (Participants) | 1200 | 1201 | 1799 | 4200
Age, Customized [Count of Participants; unit: Participants]
  18-24 | 136 | 145 | 205 | 486
  25-44 | 569 | 534 | 877 | 1980
  45-64 | 453 | 461 | 648 | 1562
  65+ | 40 | 61 | 68 | 169
  Unknown | 2 | 0 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 658 | 645 | 998 | 2301
  Male | 542 | 556 | 801 | 1899
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 638 | 609 | 888 | 2135
  Black | 191 | 194 | 307 | 692
  Hispanic | 250 | 270 | 421 | 941
  Asian | 24 | 36 | 46 | 106
  American Indian | 18 | 16 | 24 | 58
  Multi-Race | 76 | 73 | 103 | 252
  Unknown | 3 | 3 | 10 | 16
Education [Count of Participants; unit: Participants]
  <12 | 314 | 288 | 444 | 1046
  HS Diploma | 405 | 378 | 595 | 1378
  Some College | 396 | 442 | 631 | 1469
  BA/BS or Higher | 84 | 92 | 128 | 304
  Unknown | 1 | 1 | 1 | 3
Language [Count of Participants; unit: Participants]
  English | 1068 | 1049 | 1559 | 3676
  Spanish | 132 | 152 | 240 | 524
Smoke Level [Count of Participants; unit: Participants]
  6-10 | 352 | 353 | 527 | 1232
  11+ | 848 | 848 | 1272 | 2968

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Six-month Continuous Abstinence From Cigarettes
Time Frame: 7 months post enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Patch (Placebo) | Patch (Real)
Number analyzed (Participants) | 1200 | 1201 | 1799
Participants | 70 | 101 | 190

2. Secondary Outcome: Number of Participants Quit for 30-days at 2-months Post Enrollment
Time Frame: 2-months post enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Patch (Placebo) | Patch (Real)
Number analyzed (Participants) | 1200 | 1201 | 1799
Participants | 136 | 173 | 334

ADVERSE EVENTS:
Arm/Group | Usual Care | Patch (Placebo) | Patch (Real)
Serious Adverse Events (participants affected / at risk) | 0/1200 | 0/1201 | 0/1799
Other Adverse Events (participants affected / at risk) | 0/1200 | 0/1201 | 0/1799

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No